CLINICAL TRIAL: NCT05865717
Title: Exploring Determinants of Lifestyle Practices With Chronic Diseases Among Different Professionals in Islamabad Capital Territory: A Mixed Method Study
Brief Title: Lifestyle Practices With Chronic Diseases Among Different Professionals
Status: Completed | Type: Observational
Sponsor: Health Services Academy, Islamabad, Pakistan (Other)
Responsible Party: Principal Investigator, Hassan Mumtaz, Senior Clinical Research Associate, Principal Investigator, Public Health Scholar, Health Services Academy, Islamabad, Pakistan
Other Study IDs: 000223/HSA/MSPH-2021
Record Dates: First submitted 2023-03-07; First posted 2023-05-19 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Chronic Diseases in Adolescence; Cardio Vascular Disease; Diabetes Type 2
Keywords: Sedentary Professionals; Lifestyle Practices; Lifestyle Medicine; medical anthropology
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Teachers: A professional whose teaching at an academic institution from the past 3 years. e.g College or university
  Interventions: Behavioral: Quantitative sampling; Other: Qualitative interviews
- Bankers: A professional who has a desk job of at least 8-10 hours per day working in the corporate sector.
  Interventions: Behavioral: Quantitative sampling; Other: Qualitative interviews
- IT experts: A person who uses computers for work or communication, having a desk job of at least 8-10 hours per day
  Interventions: Behavioral: Quantitative sampling; Other: Qualitative interviews
- Doctors: Physicians having a desk job in their outpatient clinic for at least 8-10 hours per day
  Interventions: Behavioral: Quantitative sampling; Other: Qualitative interviews
- Administrative job personal: Personals working in the human resource department or administration department whose job involves desk work 10 hours per day.
  Interventions: Behavioral: Quantitative sampling; Other: Qualitative interviews

INTERVENTIONS:
Behavioral: Quantitative sampling — A questionnaire asks about demographics, lifestyle (including cigarette smoking) & desk job hours, eating habits, sleep patterns, mental health, and motivation. Data on the frequency and size of regular food consumption will be gathered by completing a survey. Physical activity will be measured using a questionnaire developed by the American College of Lifestyle Medicine and Loma Linda University (Lifestyle Assessment Short Form, 2018).
Other: Qualitative interviews — Thematic analysis will be done dividing into 4 different themes Personal life, professional life, Concept of Healthiness, Improving Lifestyle

SUMMARY:
A qualitative study conducted in 2018 Exploring socio-cultural factors impacting adherence to type 2 diabetes therapy in rural Sargodha featured respondents who were primarily doctors, patients, and. Diet, exercise, and smoking were all variables. The void we investigators will fill will be comprised of several professionals assessing sleep and sedentary lifestyle. A book on anthropology published in 2021 shows the gap are still the same about sedentary life style.

The investigators aim to determine lifestyle practices in relation to sedentary behaviour in different occupations & comparing which profession is prone to chronic diseases in accordance to lifestyle practices

DETAILED DESCRIPTION:
Considering all the numerous variables that can have an effect on someone's health, it seems obvious that prior research into all the potential determinants of a health intervention's success is necessary. Care for a sickness requires knowledge of both the disease itself and the patient's social and cultural context, thus it's important to learn about both. Since diabetes is chronic, it must be managed permanently. IDF's most recent projections for 2019 show that the prevalence of diabetes in Pakistan has risen dramatically. There will be 33 million diabetic adults in Pakistan in 2021, a 70% rise from 2019. After China (with 141 million cases) and India (with 102 million), Pakistan presently has the third-highest rate of diabetes prevalence worldwide (74 million). The growth in the prevalence of type 2 diabetes can be attributed to multiple variables, including but not limited to those in the areas of economics, demography, ecology, and heredity. Urbanization, an ageing population, a decline in physical activity, and a rise in overweight and obesity are all contributing factors.

In addition to providing useful information for larger-scale diabetes initiatives at the national and provincial levels (and their partners), this study's unique emphasis on the patient's point of view could be seen as groundbreaking (as an illness). The recommended treatment will be interpreted from patient's viewpoint and their respective issues, concerns, challenges and socio-cultural elements at large that may influence or compromise the adherence towards the proposed treatment of diabetes. Therefore, from the patient's vantage point, the proposed treatment's implementation through pilot intervention in chosen health facilities can be understood as an explanatory model of sickness (of/for diabetes).

ELIGIBILITY:
Inclusion Criteria:

* People between the ages of 30 and 50
* Sedentary professions, such as teachers and bankers, IT experts, doctors, administrative job personal
* Working for the past 03 years .

Exclusion Criteria:

* Disabled people who cannot move or engage in an active lifestyle .
* Those individuals already diagnosed with mental health issues

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study will be conducted using multi locale within Islamabad capital territory, including sedentary professionals, such as teachers and bankers, IT experts, doctors & administrative job personal of Islamabad, Pakistan.
  Data would be taken from the sedentary professionals, such as teachers, bankers, IT experts, doctors & administrative job personal via self-administered questionnaire through Google Forms.
Sampling Method: Probability Sample
Enrollment: 357 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Physical activity which will be measured using a questionnaire developed by the American College of Lifestyle Medicine and Loma Linda University | 04 months
  With relation to sedentary behavior in different occupations

SECONDARY OUTCOMES:
Prevalence of Chronic Diseases according to each profession and BMI | 04 months
  comparing which profession is prone to chronic diseases in accordance to lifestyle practices

CONTACTS AND LOCATIONS:
Locations (1):
- Health Services Academy, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Achievements in Public Health, 1900-1999: Changes in the Public Health System. (1999). Centers for Disease Control and Prevention.
- [Background] Khan, S. E. (2020). Exploring socio-cultural factors influencing adherence to the treatment of type 2 diabetes in rural Sargodha. Quaid-i-Azam University, Islamabad
- [Background] Khan, S. E. (2021). Life Style Change An Anthropological Perspective (1st ed.). ferozsons
- [Background] Stierlin AS, De Lepeleere S, Cardon G, Dargent-Molina P, Hoffmann B, Murphy MH, Kennedy A, O'Donoghue G, Chastin SF, De Craemer M; DEDIPAC consortium. A systematic review of determinants of sedentary behaviour in youth: a DEDIPAC-study. Int J Behav Nutr Phys Act. 2015 Oct 9;12:133. doi: 10.1186/s12966-015-0291-4. PMID 26453175
- [Background] Gonzalez K, Fuentes J, Marquez JL. Physical Inactivity, Sedentary Behavior and Chronic Diseases. Korean J Fam Med. 2017 May;38(3):111-115. doi: 10.4082/kjfm.2017.38.3.111. Epub 2017 May 23. PMID 28572885